# Statistical Analysis Plan



# **Approvals**

| Role Signatures | |
|---|---|
| | Print Name: |
| | Sign Name: |
| Biostatistician | DocuSigned by: Signer Name: Signing Reason: I am the author of this document Signing Time: 05-Jun-2023 12:16:06 EDT 02E00F9EBE524D61BC8DB1C6A31917A4 |
| | Print Name: |
| | Sign Name: |
| Peer Reviewer | DocuSigned by: Signer Name: Signing Reason: I have reviewed this document Signing Time: 05-Jun-2023 12:16:51 EDT ED5BA58B854A40FCBC2009EA1722388A |



| Role | Signatures |
|---|---|
| | Print Name: |
| | Sign Name: |
| Kimberly-Clark<br>Corporation<br>Representative | DocuSigned by: Signer Name: Signing Reason: I approve this document Signing Time: 05-Jun-2023 09:23:02 PDT CFE9F8C8EF284DCC8AB892DB97BB3DCC |

# **Document History**

| Version | Date | Author | Description |
|---|---|---|---|
| 1.0 | 15NOV2022 | | Final SAP |
| 1.1 | 03MAR2023 | | Final SAP with Amendment: 1) Updated table 14.2.2.1 by adding number of tampons remaining white and any flow. 2) Updated table 14.2.2.2 by adding reasons why subjects were not able to insert the tampon using the applicator. 3) Added listing 16.2.6.2.3 for reasons why subjects were not able to insert the tampon using the applicator 4) Updated section 8.2 and 13.4 for the updates specified above. 5) Added hypothesis testing for significant difference between treatment groups to section 8.1 and 8.2 6) Added block of difference between test and reference articles for elongation and proportion of subject who were able to insert each tampon to Table 14.2.1 and 14.2.2.2 7) Added definition of Ns to table shells. |





# **Table of Contents**

| Tal | | History | 3 |
|---|---|---|---|
| | .160 | | 5 |
| т . | oie oi C | ontents | 4 |
| L <sub>1</sub> S | t of Tab | oles | 6 |
| Lis | t of Fig | ures | 6 |
| Lis | t of Ab | previations | 7 |
| 1. | Ov | erview | 8 |
| 2. | Stu | dy Objectives and Endpoints | 8 |
| | 2.1. | Study Objective | 8 |
| | 2.1.1. | Primary Objective | 8 |
| | 2.2. | Study Endpoints | 9 |
| | 2.2.1. | Validation Criteria Endpoints | 9 |
| | 2.2.2. | Safety Endpoints | 9 |
| 3. | Ov | erall Study Design and Plan | 9 |
| | 3.1. | Overall Design | 9 |
| | 3.2. | Sample Size and Power | 10 |
| | 3.3. | Study Population | 10 |
| | 3.4. | Test Articles Administered | 11 |
| | 3.5. | Method of Assigning Subjects to Treatment Groups | 11 |
| | 3.6. | Blinding and Unblinding. | 11 |
| | 3.7. | Schedule of Events | 11 |
| 4. | Sta | tistical Analysis and Reporting | 13 |
| | 4.1. | Introduction | 13 |
| | 4.2. | Interim Analysis and Data Monitoring | 13 |
| 5. | An | alysis Populations | 13 |
| 6. | Ge | neral Issues for Statistical Analysis | 14 |
| | 6.1. | Statistical Definitions and Algorithms | 14 |
| | 6.1.1. | Handling of Dropouts or Missing Data | 14 |
| | 6.1.2. | Analysis Visit Windows | 14 |
| | 6.1.3. | Pooling of Sites | 14 |
| | 6.1.4. | Derived Variables | 14 |
| | 6.1.5. | Data Adjustments/Handling/Conventions | 14 |
| 7. | Stu | dy Subjects and Demographics | 15 |



| | 7.1. | Disposition of Subjects and Withdrawals | 15 |
|-----|--------|-------------------------------------------------|----|
| | 7.2. | Protocol Violations and Deviations | 15 |
| | 7.3. | Demographics and Other Baseline Characteristics | 16 |
| | 7.4. | Exposure and Compliance | 16 |
| 8. | Val | lidation Criteria Analysis | 16 |
| | 8.1. | Elongation | 16 |
| | 8.2. | Diary Responses | 17 |
| | 8.3. | Packaging and Labeling Interview Responses | 17 |
| | 8.4. | Product Tolerability | 18 |
| 9. | Saf | ety and Tolerability Analysis | 18 |
| | 9.1. | Adverse Events | 18 |
| | 9.1.1. | Serious Adverse Events | 19 |
| | 9.2. | Clinical Laboratory Evaluations | 19 |
| | 9.3. | Vital Signs | 20 |
| | 9.4. | Electrocardiograms | 20 |
| | 9.5. | Gynecological Examination | 20 |
| | 9.6. | Concomitant Medication | 20 |
| | 9.7. | Product Complaints | 20 |
| 10. | Cha | anges from Planned Analysis | 20 |
| 11. | Oth | ner Planned Analysis | 20 |
| | 11.1. | Coronavirus 2019 (COVID-19) Impact | 21 |
| 12. | Ret | ferences | 21 |
| 13. | Tal | bles, Listings, and Figures | 22 |
| | 13.1. | Demographic Data Summary Tables and Figures | 22 |
| | 13.2. | Validation Criteria Data | 22 |
| | 13.3. | Safety and Tolerability Data | 22 |
| | 13.4. | Planned Listing Descriptions | 24 |
| 14. | Tal | bles and Listings Shells | 26 |
| | 14.1. | Standard Layout for all Tables and Listings | 26 |
| | 14.2. | Planned Table Shells | |
| | 14.3. | Planned Listing Shells. | 52 |



# **List of Tables**

| Table 1: Schedule of Events | 12 |
|------------------------------------------------------|----|
| Table 2: Demographic Data Summary Tables and Figures | 22 |
| Table 3: Validation Criteria Data | 22 |
| Table 4: Safety and Tolerability Data | 22 |
| Table 5: Planned Listings | 24 |
| List of Figures | |
| Figure 1: Standardized Layout | 27 |
| Figure 2: Planned Table Shells | 29 |
| Figure 3: Planned Listing Shells | 53 |



# **List of Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | adverse event |
| ASA | American Statistical Association |
| ATC | anatomical therapeutic chemical |
| CI | confidence interval |
| CRF | case report form |
| CSR | clinical study report |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| ICH | International Conference on Harmonization |
| ITT | intent-to-treat |
| MedDRA | medical dictionary for regulatory activities |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SOC | system organ class |
| TSS | toxic shock syndrome |
| WHO-DD | World Health Organization drug dictionary |

#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Kimberly-Clark Corporation protocol number AFC-21-001 (An Open-Label Clinical Validation Study of an Applicator Tampon), dated 24-Aug-2022, Version 2.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials (ICH, 1998). All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA, 2018) and the Royal Statistical Society (RSS, 2014), for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be approved before any inferential or descriptive analysis of data pertaining to Kimberly-Clark Corporation's study AFC-21-001.

#### 2. Study Objectives and Endpoints

#### 2.1. Study Objective

#### 2.1.1. Primary Objective

The primary objective of this study is to validate that changes in the design of the tampons meet defined user needs. The primary objective will have been met if the following criteria are met:

- Test tampon elongation rate is the same as or better than the reference tampon for each absorbency, where same is defined as test tampon elongation rate ≤ reference tampon elongation rate.
- Product tolerability is deemed to be acceptable based on review of the results.
- Diary responses have ≥ 96% response rates consistent with each user need for each absorbency. If the rate is lower than 96%, the response rate consistent with the user need related to the test tampon must be the same as or better than the response rate of the reference tampon, where same is defined as test tampon response rate ≥ reference tampon response rate.



• Interview responses demonstrate that 95% of users are able to identify key information on the package and insert, and able to distinguish between absorbency levels on the wrappers.

#### 2.2. Study Endpoints

#### 2.2.1. Validation Criteria Endpoints

#### 2.2.1.1. Primary Endpoint

The proportion of used tampons that have elongated will be used to assess the following user need:

• User can remove product from the vagina after use

#### 2.2.1.2. Key Secondary Endpoints

The key secondary endpoints of this study include the following:

- Diary responses will be used to assess the following user needs:
  - o Product to remain clean prior to use
  - Product to remain in working condition prior to use
  - User can access the product
  - User can vaginally insert and place the tampon
  - User can remove product from the vagina after use
  - Product absorbs fluid
- Interview responses will be used to assess the following user needs:
  - User is able to distinguish between absorbency levels
  - Packaging is labeled properly
- Product tolerability will be evaluated through the following measures:
  - Gynecological exam findings
  - o Frequency and severity of adverse events

#### 2.2.2. Safety Endpoints

The safety endpoints for this study, gynecological exam findings and frequency and severity of adverse events, are included as key secondary endpoints.

#### 3. Overall Study Design and Plan

#### 3.1. Overall Design

This study is an open-label, randomized, crossover study designed to validate that changes to the design of tampons meet defined user needs. Subjects will be assigned to either a regular absorbency arm or super absorbency arm. Subjects will test a new tampon design (test tampon) and a commercially available tampon design (reference tampon).



Each tampon type will be used over the course of one menstrual cycle. Within each absorbency arm, subjects will be randomized to the order in which to use the test tampon and the reference tampon. Subject participation in the study will last over the course of 2 menstrual cycles, or approximately 2 months.

A subset of 120 subjects (60 subjects within each absorbency arm) will undergo gynecological examinations prior to and following tampon use. For the subset of subjects undergoing gynecological exams, the study will include a total of 4 visits, 2 visits for each menstrual cycle. The first visit will be the screening visit and the first pre-use visit. The next visit will be the first post-use visit, followed by the second pre-use visit and the second post-use visit. Pre-use visits will be conducted within 72 hours prior to expected menstruation and post-use visits will be conducted within 72 hours following the last tampon use for that menstrual cycle. Gynecological examinations will be performed at each visit. This subset of subjects will also complete a packaging and labeling interview at the first visit to assess whether subjects can identify and distinguish key information on the product packaging.

For the remainder of subjects who will not undergo gynecological examinations, the study will include 3 visits: a screening/pre-use visit and 2 post-use visits. Post-use visits will be conducted within 72 hours following the last tampon use for that menstrual cycle.

All subjects will keep a diary during menstruation with entries for each tampon used and will collect each used tampon to be returned to the site. At each post-use visit, site personnel will review subject diaries for completeness and accuracy, record the number of used and unused tampons returned, and evaluate used tampons to assess tampon integrity. Subjects will be considered to have completed the study after they complete the second post-use visit. Refer to the Schedule of Events (Table 1) for more details.

#### 3.2. Sample Size and Power

The sample size was calculated for a single absorbency and is based on the assumption that 0.7% of reference tampons elongate (>10 mm) upon removal and 0.2% of test tampons elongate upon removal. An estimated yield of 43.75% was used, where yield is the number of usable tampons for the elongation analysis divided by the total number of products given to the subjects (i.e., yield means the percentage of tampons given to each subject that were used and can be included in the elongation analysis). It is assumed that subjects are given 16 reference tampons and 16 test tampons and use 7 tampons in each cycle.

With a power of 80% and a 2-sided alpha of 0.05, assuming 2 tampon types tested (reference and test) and each subject receiving 16 products per cycle, a total of 369 subjects will need to be enrolled in the study for each absorbency. Since there are 2 absorbencies, the study will enroll 738 subjects.

For each absorbency this translates into needing a total of 5,166 used tampons (2,538 used tampons for each tampon type (reference and test)).

#### 3.3. Study Population

The study population consists of female subjects, ages 18-49, in good general health, in the AD-ST-33.06 Effective date: 12-Nov-2020



United States who normally use tampons for menstrual protection, menstruate regularly, and do not have a history of Toxic Shock Syndrome (TSS).

#### 3.4. Test Articles Administered

Subjects will be assigned to one of two arms in the study based on the absorbency of tampon the subject uses most often: a regular absorbency arm or a super absorbency arm. Within each arm, subjects will be randomly assigned to the order in which to test a new, modified tampon design (test tampon) and a currently marketed, commercial tampon (reference tampon). Each tampon, test or reference, will be administered for use over the course of one menstrual cycle. Subjects will be administered a box with 16 tampons per menstrual cycle. The test article codes are listed below.

| Test Article Description | <b>Test Article Code</b> |
|---|---|
| Modified Tampons (test tampons) – regular absorbency | BR |
| Commercial Tampons (reference tampons) – regular absorbency | CR |
| Modified Tampons (test tampons) – super absorbency | BS |
| Commercial Tampons (reference tampons) – super absorbency | CS |

#### 3.5. Method of Assigning Subjects to Treatment Groups

Subjects will be assigned a unique subject identification number by the site at screening. Following completion of screening procedures, eligible subjects will be assigned to either the regular or super absorbency arm, based on the tampon absorbency the subject uses most often. Within each arm, the order in which the test and reference tampons will be used will be randomized.

A randomization schedule that was created by a biostatistician at will be provided to each site. Blinding was not required as this is an open-label study. Unique subject randomization numbers will be assigned by the site according to the site-specific randomization schedule. Randomization numbers should be assigned sequentially within each arm.

### 3.6. Blinding and Unblinding

Not applicable as this is an open-label study.

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1.



# **Table 1: Schedule of Events**

| Event | Visit 1<br>Screening/Baseline | Visit 2<br>Post-Use Visit | Visit 3<br>Pre-Use Visit | Visit 4<br>Post-Use Visit | Unscheduled<br>Visit |
|---|---|---|---|---|---|
| Informed Consent | х | | | | |
| Inclusion/Exclusion | х | | | | |
| Demographics | х | | | | |
| Medical History | х | | | | |
| Concomitant Medications | Х | Х | Х | Х | Х |
| Gynecological Symptom<br>Assessment | х | Х | Х | Х | Х |
| Gynecological Exam<br>(Visual inspection, infection<br>assessment, vaginal discharge,<br>and vaginal pH) | Х | Х | Х | Х | Х |
| Packaging/Labeling Interview | X | | | | |
| Randomization | Х | | | | |
| Test Article and Diary<br>Dispensation | Х | X* | X* | | |
| Diary Training | X | X* | X* | | |
| Test Article Collection<br>(Used and unused products) | | Х | | Х | |
| Diary Review | | Х | | Х | |
| Tampon Integrity Assessment | | Х | | Х | |
| Adverse Event Collection | | Х | Х | Х | Х |
| Study Completion | | | | Х | |

<sup>\*</sup>As needed

Key:

| Х | Conducted for all subjects |
|---|---|
| X | Conducted for a subset of 120 subjects (Note, visit 3 is only required for this subset of subjects) |

### 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing and tabulation of descriptive statistics described in this SAP will primarily use SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. Summaries may include 95% confidence intervals (CIs) if appropriate. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population, either overall or within each absorbency arm, unless otherwise specified.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data. Measures of spread (SD, 95% CI) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified. General exceptions to this rule are values of 100% which will be displayed without any decimal places and zero counts which will not display percentages.

No inferential statistical hypothesis testing will be performed to assess whether the validation criteria have been met. All the analyses described in this SAP to assess whether validation criteria have been met are descriptive.

#### 4.2. Interim Analysis and Data Monitoring

No interim analyses are planned.

#### 5. Analysis Populations

The following analysis populations are planned for this study:

- Intent-To-Treat Population (ITT): The ITT population includes all subjects randomized into the study.
- **Safety Population:** The Safety Population includes all ITT subjects who insert at least 1 tampon.
- Modified Intent-To-Treat Population (MITT): The MITT population includes all safety subjects who have no major protocol deviations and return at least 1 tampon that can be assessed for elongation.



Assignment of subjects to populations will be determined at a data review meeting prior to database lock.

#### 6. General Issues for Statistical Analysis

#### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Handling of Dropouts or Missing Data

In general, missing data will not be imputed unless otherwise stated.

#### 6.1.2. Analysis Visit Windows

Analysis visits will be assigned based on the nominal visit recorded in the study database.

#### **6.1.3.** Pooling of Sites

Data will be pooled across sites for analysis.

#### 6.1.4. Derived Variables

• Elongated = Any used tampon with a measurement of elongation >10 mm will be considered elongated.

#### 6.1.5. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA; version 25.1) thesaurus. Concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD) Enhanced B3 (September 2022).

The first article insertion date will be the date of the first tampon insertion, that the subject reported, but only for a tampon that has both the date of the tampon's insertion and the date of the tampon's removal documented in the diary. The last article's removal date will be defined in the same manner. The first insertion and last removal dates within each menstrual cycle will be identified using a similar logic but using the data from each menstrual cycle.

In case the subject didn't report the tampon's insertion and removal dates for the 1st menstrual period in the diary but returned at least 1 used tampon from 1st menstrual cycle and has available diary data for the 2nd menstrual cycle, then the first article insertion date and last article removal date for the 1st menstrual cycle will be calculated from the date of post-use visit 2 with the



assumption, that number of days between first tampon's insertion and post-use visits are the same for both menstrual cycles.

If partial adverse event onset dates or partial medication dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows: if just day is missing then the day assigned is the first day of the month or the date of first test article insertion (if in the same month), whichever is later; if just month is missing then the month assigned is the month of the first test article insertion, unless that results in a date before the first test article insertion in which case the month after the first test article insertion is used; and if both month and day are missing then the month assigned is the month of the first test article insertion and the day assigned is either the first day of the month or the first test article insertion date, whichever is later.

If partial adverse event onset times occur, the convention is as follows: if the missing time occurs on the day of the first test article insertion and both the hour and minute are missing then the time assigned is the time of the first test article insertion, otherwise if both the hour and minute are missing and the date is not the date of first test article insertion the time assigned is 12:00; if the date is the same as the date of the first test article insertion and only hour is missing the hour assigned is 12 or the hour of first test article insertion, whichever is later, and if the date is the same as the date of first test article insertion and only the minute is missing the minute assigned is 30 or the minute of first test article insertion, whichever is later. Otherwise the hour assigned is 12 if the hour is missing and the date is not the same as the date of first test article insertion and the minute assigned is 30 if the the date is not the same as the date of first test article insertion.

The following precatution will be considered when applying these conventions to adverse event onset dates and times: if the missing date and time reflect the date and time of onset of an adverse event, the modified date and time will be constructed to match the first documented date/time post test article administration while preserving the order in which the adverse event (AE) was reported in the CRF.

#### 7. Study Subjects and Demographics

#### 7.1. Disposition of Subjects and Withdrawals

The number of subjects randomized, the number of subjects completing, the number of subjects who withdraw early (including tabulated reasons for discontinuation from the study), and the number of subjects in each analysis population will be tabulated by absorbency arm and overall.

#### 7.2. Protocol Violations and Deviations

Protocol deviations will be classified as minor or major and will be presented in a data listing.



### 7.3. Demographics and Other Baseline Characteristics

Demographic variables such as age, sex, race, and ethnicity will be summarized overall and by absorbency arm. Baseline characteristics such as the number of tampons typically used during period and the tampon absorbency used most often will also be summarized.

Demographic and baseline characteristic data will be summarized by absorbency arm and overall for the ITT population.

#### 7.4. Exposure and Compliance

The number of used and unused tampons returned and the frequency and percentage of diaries returned with an entry present for each used tampon will be summarized by absorbency arm and overall for the Safety population.

Test article and diary dispensation information and diary review information will be listed.

#### 8. Validation Criteria Analysis

All the analyses performed to assess whether validation criteria have been met will be performed separately for each absorbency arm, with the exception of the analysis of the packaging and labeling interview responses which will be analyzed for both absorbencies combined.

#### 8.1. Elongation

Descriptive statistics will be reported for the length of elongation of used tampons within each test article type (test or reference tampon), and separately for each absorbency arm, in the MITT population. The number and percentage of used tampons that have elongated will be reported for test tampons and reference tampons. Determination of whether a tampon is considered to have elongated is described in Section 6.1.4. The denominator for the percentage calculation will be based upon the number of used tampons returned within each test article type (test or reference tampon) and within each absorbency arm (regular or super). The 95% CIs for the percentage elongated estimates will be computed using the exact method (Clopper & Pearson, 1934).

In addition, the testing of equality of proportions of elongation between test and reference article types within each absorbency arm will be performed. For this purpose, the difference between proportions will be calculated along with 95% Wald CIs. Pearson chi-square test will be computed in support of hypothesis testing. The samples for comparison will be considered independent.

The following hypothesis will be tested:

H0: p1-p2=0. There is no significant difference in the tampon's elongation rate between the test and reference article types within each absorbency arm.

H1:  $p1-p2\neq0$ . There is a significant difference in the tampon's elongation rate between the test and reference article types within each absorbency arm.

#### 8.2. Diary Responses

The number and percentage of diary responses will be reported for test tampon diary entries and reference tampon diary entries in the Safety population, and separately for each absorbency arm. Diary responses for individual tampon entries will be summarized separately from diary responses following last tampon use. Diary responses for individual tampon entries were reported specific to each tampon used and were recorded repeatedly for each used tampon throughout a given menstrual cycle. The denominator for the percentage calculation for individual tampon entry diary responses will be based upon the total number of used tampon diary entries within each question and within each test article type and within each absorbency arm. The number of tampons remaining white and when the subject reported having any flow when using the tampon will be summarized within each test article type and within each absorbency arm as well. The denominator for the percentage calculation will be the total number of used tampon diary entries within each question and within each test article type and within each absorbency arm. Diary responses recorded following last tampon use were reported only once per menstrual cycle. The reasons for not inserting the tampon using the applicator will be summarized. The denominator for the percentage calculation for diary responses following last tampon use will be based on the total number of diary entries within each question and within each test article type and within each absorbency arm. Individual diary responses and diary responses recorded following the last tampon will be listed. And additionally, the reasons for not inserting the tampon using the applicator will be presented in a separate listing. The 95% CIs for the percentage of patients who are able to insert each tampon will be computed using the exact method (Clopper & Pearson, 1934).

In addition, the testing of equality of proportions of patients who are able to insert each tampon between test and reference article types within each absorbency arm will be performed. For this purpose, the difference between proportions will be calculated along with 95% Wald CIs. Pearson chi-square test will be computed in support of hypothesis testing. The samples for comparison will be considered independent.

The following hypothesis will be tested:

H0: p1-p2=0. There is no significant difference in proportions of patients who are able to insert each tampon between the test and reference article types within each absorbency arm.

H1:  $p1-p2\neq0$ . There is a significant difference in proportions of patients who are able to insert each tampon between the test and reference article types within each absorbency arm.

### 8.3. Packaging and Labeling Interview Responses

The packaging and labeling interview will be administered at the Screening/Baseline Visit (Visit 1) to the subset of subjects who were selected to undergo gynecological exams prior to and following tampon use. The number and percentage of subjects that were able to correctly identify and distinguish key product information will be reported for the subset of subjects in the ITT population who undergo gynecological examinations and complete the packaging and labeling interview. A subject will be considered to have correctly identified the information if they: 1)



correctly identify the key product information in their first response, or 2) correctly identify the information after a follow-up question from the interviewer. The summary will be presented for the subset of subjects in the ITT population overall, not by absorbency arm. The denominator for the percentage calculation will be based upon the total number of subjects in the ITT population who belong to the subset of subjects that were selected to undergo gynecological exams and complete the packaging and labeling interview.

#### 8.4. Product Tolerability

Product tolerability will be evaluated through gynecological exam findings and frequency and severity of adverse events. The analysis of adverse events is presented in Section 9.1 and the analysis of gynecological exam findings is presented in Section 9.5.

### 9. Safety and Tolerability Analysis

Safety and tolerability will be evaluated from reported adverse events (AEs) and gynecological exam findings. All safety analyses will be performed on the Safety population. Analyses will be performed separately for each absorbency arm.

#### 9.1. Adverse Events

All AEs and serious adverse events (SAEs) will be coded using the MedDRA v. 25.1.

All AE data will be summarized for 3 periods: before any test article use, during and following test tampon use, during and following reference tampon use. AEs will be assigned to an analysis period based on the below criteria. The criteria for assigning AEs to an analysis period will differ depending on the type of test article (reference or test tampon) first used by the subject.

| Test article order | Criteria for assigning AEs to analysis periods |
|---|---|
| Reference tampon → Test tampon | If the start date of the adverse event was before the date of first insertion of a reference tampon, then the AE will be assigned to the "before any test article use" period. |
| | If the start date of the adverse event was on or after<br>the date of first insertion of a reference tampon, but<br>before the date of first insertion of a test tampon, then<br>the adverse event will be assigned to the "during and<br>following reference tampon use" period. |
| | If the start date of the adverse event was on or after<br>the date of first insertion of a test tampon, then the<br>adverse event will be assigned to the "during and<br>following test tampon use" period. |



# Test tampon → Reference tampon

If the start date of the adverse event was before the date of first insertion of a test tampon, then the AE will be assigned to the "before any test article use" period.

If the start date of the adverse event was on or after the date of first insertion of a test tampon, but before the date of first insertion of a reference tampon, then the adverse event will be assigned to the "during and following test tampon use" period.

If the start date of the adverse event was on or after the date of first insertion of a reference tampon, then the adverse event will be assigned to the "during and following reference tampon use" period.

An overall summary of AEs will be provided; this will present number and percentage of subjects who reported at least 1 of the following: any AE, AEs by maximum severity, AEs by maximum relationship to study product, AEs by maximum frequency, and SAEs.

In addition to the overall summary, summaries of the number and percentage of subjects with AEs will be displayed for each absorbency arm, grouped by MedDRA system organ class and preferred term (coded using MedDRA v. 25.1). Summaries of AEs by severity, relationship to study product, and frequency will also be provided. In the case of multiple occurrences of the same AE within the same subject, each subject will only be counted once for each preferred term.

In the summaries showing severity, relationship to study product, and frequency, the event with the maximum severity, strongest relationship, and highest frequency, respectively, will be reported. If a particular event is missing the severity, relationship, or frequency then the strongest possible severity, relationship, or frequency will be assumed for analysis (severity = severe, relationship = definitely related, frequency = continuous).

A data listing of all AEs will be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.1. Serious Adverse Events

All SAEs that occur during the study will be listed by absorbency arm and also tabulated by system organ class and preferred term and presented by absorbency arm.

#### 9.2. **Clinical Laboratory Evaluations**

No clinical laboratory evaluations are planned to be collected for this study.

#### 9.3. Vital Signs

No vital signs are planned to be collected for this study.

#### 9.4. Electrocardiograms

No electrocardiograms are planned to be performed for this study.

#### 9.5. Gynecological Examination

A subset of subjects will undergo a gynecological examination at each study visit prior to and following tampon use. Vaginal pH, and the number and percentage of subjects with any lesions, a suspected infection, other abnormal findings, and a clinically significant result will be summarized separately for each absorbency arm using the subset of subjects in the Safety population who underwent gynecological examinations. Complete gynecological examination information will be listed.

#### 9.6. Concomitant Medication

Medications will be coded using World Health Organization Drug Dictionary (WHO-DD) Enhanced B3 (September 2022).

All medication data will be listed. The listing will indicate whether the medication is considered a prior medication, concomitant medication, or both. Medications that started before first test article insertion date will be considered prior medications whether or not they were stopped before first test article insertion date. Any medications continuing or starting after first test article insertion date will be considered to be concomitant. If a medication starts before first test article insertion date and continues after first test article insertion date it will be considered both prior and concomitant.

#### 9.7. Product Complaints

Information on product complaints that were not captured in the subject diaries or as adverse events will be provided in a separate listing.

#### 10. Changes from Planned Analysis

Not applicable.

#### 11. Other Planned Analysis

Not applicable.



### 11.1. Coronavirus 2019 (COVID-19) Impact

Should a study visit be affected by COVID-19, study staff will record how the visit was affected. This information will be presented in a listing.

#### 12. References

ASA. (2018) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2018. <a href="http://www.amstat.org/about/ethicalguidelines.cfm">http://www.amstat.org/about/ethicalguidelines.cfm</a>

Clopper, C. J., & Pearson, E. S. (1934). The use of confidence or fiducial limits illustrated in the case of the binomial. *Biometrika*, 26(4), 404-413.

ICH (1998). ICH Harmonised Tripartite Guideline. Statistical Principles for Clinical Trials E9; 1998. https://database.ich.org/sites/default/files/E9\_Guideline.pdf

RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. https://rss.org.uk/about/policy-and-guidelines/code-of-conduct/.

AD-ST-33.06 Effective date: 12-Nov-2020

Version Final 1.1 | Date 05-Jun-2023 | AD-PR-109.02 Effective date: 17-Aug-2020 Page 21 of 73



### 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (e.g., listing number).

The following are planned summary tables for protocol number AFC-21-001. The table numbers and page numbers are place holders only and will be determined when the tables are produced.

#### 13.1. Demographic Data Summary Tables and Figures

Table 2: Demographic Data Summary Tables and Figures

| Table Number | Population | Table Title / Summary |
|--------------|--------------|-------------------------------------------|
| Table 14.1.1 | All subjects | Subject Disposition |
| Table 14.1.2 | ITT | Demographics and Baseline Characteristics |
| Table 14.1.3 | Safety | Exposure to Study Product |

#### 13.2. Validation Criteria Data

**Table 3: Validation Criteria Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.2.1 | MITT | Summary of Elongated Tampons |
| Table 14.2.2.1 | Safety | Summary of Individual Tampon Entry Diary Reponses |
| Table 14.2.2.2 | Safety | Summary of Diary Responses Following Last Tampon Use |
| Table 14.2.3 | ITT, Gynecological<br>Exam Subset | Summary of Packaging and Labeling Interview Responses |

#### 13.3. Safety and Tolerability Data

**Table 4: Safety and Tolerability Data** 

| Table Number | Population | Table Title / Summary |
|---|---|---|
| 14.3.1 Displays of | f Adverse Events | |
| Table 14.3.1.1 | Safety | Overall Summary of Adverse Events |
| Table 14.3.1.2 | Safety | Adverse Events by System Organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Adverse Events by System Organ Class, Preferred Term, and Maximum Severity |



| Table Number | Population | Table Title / Summary |
|---|---|---|
| Table 14.3.1.4 | Safety | Adverse Events by System Organ Class, Preferred Term, and Maximum Relationship to Study Product |
| Table 14.3.1.5 | Safety | Adverse Events by System Organ Class, Preferred Term, and Maximum Frequency |
| 14.3.2 <b>Summary</b> | of Deaths, Other Seri | ous and Significant Adverse Events |
| Table 14.3.2.1 | Safety | Serious Adverse Events by System Organ Class and Preferred Term |
| 14.3.3 Narratives | of Deaths, Other Ser | ious and Certain Other Significant Adverse Events |
| Table 14.3.3.1 | e 14.3.3.1 Safety Listing of Serious Adverse Events | |
| 14.3.6 Other Safe | ety Data Summary Ta | bles |
| Table 14.3.6.1.1 | Safety,<br>Gynecological Exam<br>Subset | Gynecological Examination – Visual Assessment Details |
| Table 14.3.6.1.2 | Safety,<br>Gynecological Exam<br>Subset | Gynecological Examination – Additional Findings |





## 13.4. Planned Listing Descriptions

The following are planned data and subject data listings for protocol number AFC-21-001.

In general, one listing will be produced per CRF domain. All listings will be sorted by absorbency arm, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed. Screen failures will only be presented in Listings 16.2.1.1, 16.2.2.1, and 16.2.2.3; otherwise, only enrolled subjects will be listed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 5: Planned Listings** 

| Listing Number | Population | Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listin | gs | |
| 16.2.1 Subject Discontin | uations/Completions | |
| Listing 16.2.1.1 | All Subjects | Subject Disposition |
| 16.2.2 Protocol Deviation | ns | |
| Listing 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria |
| Listing 16.2.2.2 | All Subjects | Protocol Deviations |
| Listing 16.2.2.3 | Screen Failures | Reason for Screen Failures |
| 16.2.3 Patients/Subjects | Excluded from the V | Validation Criteria Analyses |
| Listing 16.2.3.1 | All Subjects | Analysis Populations |
| 16.2.4 Demographic Dat | a and Other Baselin | e Characteristics |
| Listing 16.2.4.1 | All Subjects | Subject Consent and Demographics |
| Listing 16.2.4.2 | All Subjects | All Subjects Medical History |
| Listing 16.2.4.3 | All Subjects | Tampon Use Questionnaire |
| 16.2.5 Compliance Data | | |
| Listing 16.2.5.1 | All Subjects | Test Article and Diary Dispensation and Diary Training |
| Listing 16.2.5.2 | Safety Population | Diary Review |
| 16.2.6 Individual Valida | tion Criteria Data | |
| Listing 16.2.6.1 | Safety Population | Tampon Integrity Assessment |
| Listing 16.2.6.2.1 | Safety Population | Individual Tampon Entry Diary Responses |
| Listing 16.2.6.2.2 | Safety Population | Diary Responses Following Last Tampon Use |



| Listing Number | Population | Listing Title / Summary |
|---|---|---|
| 16.2 Subject Data Listin | gs | |
| Listing 16.2.6.2.3 | Safety Population | Reason for Not Inserting the Tampon Using the Applicator |
| Listing 16.2.6.3 | Gynecological<br>Exam Subset | Packaging and Labeling Interview |
| 16.2.7 Adverse Event Lis | stings (by Subject) | |
| Listing 16.2.7.1 | All Subjects | Adverse Events |
| 16.2.9 Other Clinical Ob | servations and Meas | surements (by Subject) |
| Listing 16.2.9.1.1 | Gynecological<br>Exam Subset | Gynecological Examination – Visual Assessment Details |
| Listing 16.2.9.1.2 | Gynecological<br>Exam Subset | Gynecological Examination – Additional Findings |
| Listing 16.2.9.2 | All Subjects | Prior and Concomitant Medications |
| Listing 16.2.9.3 | All Subjects | Product Complaints |
| 16.2.10 Other Study Mes | asurements or Assess | sments (by Subject) |
| Listing 16.2.10.1 | All Subjects | COVID-19 Impact Assessment |

Statistical Analysis Plan, Sponsor Kimberly-Clark Corporation Protocol Number AFC-21-001 PCN Number KIMB228084



# 14. Tables and Listings Shells

## 14.1. Standard Layout for all Tables and Listings

The following standard layout will be applied to all Tables and Listings in support of this study. Note that programming notes may be added if appropriate after each shell.

AD-ST-33.06 Effective date: 12-Nov-2020

Version Final 1.1 | Date 05-Jun-2023 | AD-PR-109.02 Effective date: 17-Aug-2020 Page 26 of 73





# Figure 1: Standardized Layout

| Kimberly-Clark Corporation | Page xx of xx |
|---|---|
| Protocol: AFC-21-001 | Version |
| <table, figure="" listing,=""> xx.x.x</table,> | |
| <title figure="" listing,="" of="" or="" table,="">&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If directly Applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 1 &lt; if applicable &gt; Recommendation is to keep footnotes to a minimum&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 2 &lt; if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n &lt; if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n+1 &lt; pgm path and name&gt;, &lt; date&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |





See Figure 2 below.





Figure 2: Planned Table Shells

Table 14.1.1 Subject Disposition All Subjects

| Status | Regular Absorbency<br>(N=XX) | Super Absorbency<br>(N=XX) | Overa <b>ll</b><br>(N=XX) |
|---|---|---|---|
| Category | (N-XX) | (N-XX) | (N-\\) |
| Screened for Eligibility | | | xx |
| Screen Failure | | | xx |
| Enrolled | XX | XX | xx |
| Randomized | xx | xx | XX |
| ITT Population [1] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gynecological Exam Subset [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Safety Population [3] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gynecological Exam Subset [2] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| MITT Population [4] | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Completed Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued Early | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrew Consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol Violation / Non-Compliance | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Investigator / Sponsor Decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to Follow-Up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Abbreviations: ITT = intent-to-treat; MITT = modified intent-to-treat.

Note: Percentages are n/Number of subjects in the ITT Population within absorbency arm and overall subjects \*100. .

<sup>[1]</sup> The ITT Population includes all subjects randomized into the study.

<sup>[2]</sup> A subset of subjects was selected to undergo gynecological exams prior to and following tampon use. In addition, only the subjects in this subset completed the packaging and labeling interview.

<sup>[3]</sup> The Safety Population includes all ITT subjects who insert at least 1 tampon.

<sup>[4]</sup> The MITT Population includes all subjects in the Safety population who have no major protocol deviations and return at least 1 tampon that can be assessed for elongation. n is the number of subjects within each category. N is the number of subjects within absorbency arm. Reference Listing: 16.2.1.1





Table 14.1.2
Demographics and Baseline Characteristics
ITT Population

| Variable | Regular Absorbency | Super Absorbency | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Age (years) [1] | | | |
| n | XX | XX | XX |
| Mean (SD) | XX,X (XX,XX) | XX.X (XX.XX) | XX X (XX XX) |
| Median | XX.X | xx x | xx x |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Gender | | | |
| Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Undifferentiated | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unknown | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| Race | | | |
| American Indian or Alaska Native | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Asian | XX (XX,X%) | XX (XX,X%) | XX (XX.X%) |
| Black or African American | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| More than One Race | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Reported | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ethnicity | | | |
| Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Hispanic or Latino | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Reported | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unknown | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ITT = intent-to-treat; SD = standard deviation.

Note: Percentages are n/Number of subjects in the ITT Population within absorbency arm and overall subjects \* 100. Demographic information including age, gender, race, and ethnicity was collected at the Screening/Baseline Visit (Visit 1). Baseline characteristics including typical tampon use were obtained at the Screening/Baseline Visit (Visit 1) from the Tampon Use Questionnaire.

[1] Age was calculated as the integer difference in years between the subject's date of informed consent and date of birth.

n is the number of subjects within each category. N is the number of subjects within absorbency arm.

Reference Listings: 16.2.4.1; 16.2.4.3





Table 14.1.2 (cont'd.)
Demographics and Baseline Characteristics
ITT Population

| Variable | Regular Absorbency | Super Absorbency | Overa <b>li</b> |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Total tampons typically used during period | | | |
| Five or less | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Six or more | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Tampon Absorbency Used Most Often | | | |
| Light | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Regular | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Super | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Super Plus | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ultra | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Equal numbers of two or more absorbencies | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX,X%) | XX (XX,X%) | XX (XX.X%) |

Abbreviations: ITT = intent-to-treat; SD = standard deviation.

Note: Percentages are n/Number of subjects in the ITT Population within absorbency arm and overall subjects \* 100. Demographic information including age, gender, race, and ethnicity was collected at the Screening/Baseline Visit (Visit 1). Baseline characteristics including typical tampon use were obtained at the Screening/Baseline Visit (Visit 1) from the Tampon Use Questionnaire.

[1] Age was calculated as the integer difference in years between the subject's date of informed consent and date of birth.

Reference Listings: 16.2.4.1; 16.2.4.3





Table 14.1.3
Exposure to Study Product
Safety Population

| Test Article Type<br>Variable | Dogular Abaarbanay | Cupar Abaarbanay | Overall |
|---|---|---|---|
| | Regular Absorbency | Super Absorbency | Overall |
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Reference Tampon | | | |
| Number of unused tampons returned | | | |
| n [1] | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Number of used tampons returned | | | |
| n [1] | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Diary entry present for each tampon used [2] | xx | xx | XX |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviation: SD = standard deviation.

Note: Percentages are n/Number of subjects, who responded to the question, in the Safety Population within absorbency arm and overall\*100. Diary review and assessment of the number of unused and used tampons returned was performed at the post-use visits which were conducted within 72 hours following the last tampon use for that menstrual cycle. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle. N is the number of subjects within each article and within absorbency arm.

[1] n is the number of tampons.

[2] n is the number of subjects, who responded to the question.

Reference Listings: 16.2.5.2; 16.2.6.1





Table 14.1.3 (cont'd.) Exposure to Study Product Safety Population

| Test Article Type Variable | Regular Absorbency | Super Absorbency | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Test Tampon | | | |
| Number of unused tampons returned | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Number of used tampons returned | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx,x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Diary entry present for each tampon used | | | |
| Yes | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviation: SD = standard deviation.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency arm and overall\*100. Diary review and assessment of the number of unused and used tampons returned was performed at the post-use visits which were conducted within 72 hours following the last tampon use for that menstrual cycle. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle.

Reference Listings: 16.2.5.2; 16.2.6.1





#### Table 14.2.1 Summary of Elongated Tampons MITT Population

| Variab <b>l</b> e | Test Tampon | Reference Tampon |
|---|---|---|
| Statistic | (N=XX) | (N=XX) |
| Length of Elongation | | |
| n [1] | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X |
| Min, Max | XX, XX | XX, $XX$ |
| Elongated [2] | | |
| n [1] | XX | XX |
| Percentage | XX.XX% | XX.XX% |
| 95% CI for the Percentage [3] | XX.XXX%, XX.XXX% | XX.XXX%, XX.XXX% |
| Difference in Percentage | XX.XX% | |
| 95% CI for the Difference in Percentage [4] | XX.XXX%, XX.XXX% | |
| Chi-Square | XX.X | |
| P-Value | X,XXX | |

Abbreviations: CI = confidence interval; MITT = modified intent-to-treat; SD = standard deviation.

Note: Percentages are n/Number of used tampons returned by subjects in the MITT Population within tampon type\*100. Length is measured in millimeters (mm). Tampon integrity assessments were performed at the post-use visits which were conducted within 72 hours following the last tampon use for that menstrual cycle. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle. N is the number of subjects within each article and within absorbency arm.

- [1] n is the number of tampons.
- [2] Any used tampon with a measurement of elongation >10 mm was considered elongated.
- [3] The 95% CIs for the percentage elongated estimates were computed using the exact method.
- [4] The 95% CIs for the difference in percentage elongated estimates were computed using Wald method

Reference Listing: 16.2.6.1

Programming Note: Repeat for Absorbency Arm: Super.



Table 14.2.2.1 Summary of Individual Tampon Entry Diary Responses Safety Population

| Variable | Test Tampon | Reference Tampon |
|---|---|---|
| Category | (N=XX) | (N=XX) |
| Able to remove the tampon | XX | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| White area remaining on tampon | XX | XX |
| No areas on the tampon remained white | XX (XX.X%) | XX (XX.X%) |
| Less than half of the tampon remained white | XX (XX.X%) | XX (XX.X%) |
| About half of the tampon remained white | XX (XX.X%) | XX (XX X%) |
| More than half of the tampon remained white | XX (XX.X%) | XX (XX.X%) |
| Whole product remained white | XX (XX.X%) | XX (XX.X%) |
| Flow when using the tampon | XX | XX |
| No flow | XX (XX.X%) | XX (XX.X%) |
| Spotting only | XX (XX.X%) | XX (XX.X%) |
| Light | XX (XX.X%) | XX (XX.X%) |
| Medium | XX (XX.X%) | XX (XX.X%) |
| Heavy | XX (XX.X%) | XX (XX.X%) |
| Tampons remaining white and where subject reported having any flow when using the tampon* | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of used tampon diary entries recorded by subjects in the Safety Population within each question and within tampon type\*100. Subject diaries were returned at the post-use visits which were conducted within 72 hours following the last tampon use for that menstrual cycle. Diary responses for individual tampon entries were reported specific to each tampon used and were recorded repeatedly for each used tampon throughout a given menstrual cycle. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle.

n is the total number of diary entries for each section of the table. N is the number of subjects within each article and within absorbency arm.

Reference Listing: 16.2.6.2.1

Programming Note: Repeat for Absorbency Arm: Super.

<sup>\*</sup>Subjects must have reported both the whole product remained white and reported anything other than "No flow". Percentages are n/Number of used tampon diary entries recorded by subjects in the Safety Population that indicate anything other than "No Flow" within tampon type\*100.



| Variable Cotonomic | Test Tampon | Reference Tampon |
|---|---|---|
| Category | (N=XX) | (N=XX) |
| Able to open the box to retrieve wrapped tampons | XX | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| 140 | XX (XX.X 70) | XX (XX.X 70) |
| Able to open each tampon wrapper | XX | XX |
| Yes | XX (XX,X%) | XX (XX,X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Fampons were clean prior to use | xx | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No. | | |
| NU | XX (XX.X%) | XX (XX.X%) |
| Able to insert each tampon using the applicator | XX | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX,X%) | XX (XX,X%) |
| Percentage of patients who are able to insert each tampon | XX.XX% | xx.xx% |
| using the applicator | | |
| 95% CI for the Percentage [1] | XX.XXX%, XX.XXX% | XX.XXX%, XX.XXX% |
| Difference in Percentage | XX.XX% | |
| 95% CI for the Difference in Percentage [1] | XX.XXX%, XX.XXX% | |
| Chi-Square | XX.X | |
| P-Value | x.xxx | |
| r-value | <b>*.</b> *** | |
| Able to insert each tampon using the applicator (diary #1) | XX | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No No | XX (XX.X%) | XX (XX.X%) |
| 110 | AA (AA.A /0) | // (//.///0) |
| Able to insert each tampon using the applicator (diary #2) | XX | XX |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Reason why was not able to insert tampon using the applicator | XX | XX |
| Not able to fully extend the applicator | XX (XX.X%) | XX (XX.X%) |
| | | /// (////////////////////////////////// |




| No tampon in the applicator | XX (XX.X%) | XX (XX.X%) |
|-----------------------------|------------|------------|
| Applicator was damaged | XX (XX.X%) | XX (XX X%) |
| Other | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of recorded diary entries by subjects in the Safety Population within each question and within tampon type\*100. Subject diaries were returned at the post-use visits which were conducted within 72 hours following the last tampon use for that menstrual cycle. Diary responses recorded following last tampon use were reported only once per menstrual cycle. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle.

n is the total number of diary entries for each section of the table. N is the number of subjects within each article and within absorbency arm.

[1] The 95% CIs for the percentage of patients who are able to insert each tampon using the applicator and for the difference in percentage of patients who are able to insert each tampon using the applicator were computed using the exact method.

Reference Listing: 16.2.6.2.2

Programming Note: Repeat for Absorbency Arm: Super.





# Table 14.2.3 Summary of Packaging and Labeling Interview Responses ITT Population Gynecological Exam Subset

| Variable | Overa <b>ll</b> |
|---|---|
| Category | (N=XX) |
| Able to correctly identify tampon absorbency provided in the regular absorbency box | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Able to correctly identify the tampon absorbency ranges for the entire line of products on the box | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Able to correctly identify the Toxic Shock Syndrome warning on the box | XX |
| Yes | XX (XX.X%) |
| No | xx (xx.x%) |
| Able to correctly identify the information that states how long you should use a tampon on the box | XX |
| Yes | XX (XX.X%) |
| No | xx (xx.x%) |
| Able to correctly identify tampon absorbency provided in the super absorbency box | XX |
| Yes | XX (XX.X%) |
| No | xx (xx.x%) |
| Able to correctly identify tampon absorbency provided in the super plus absorbency box | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |

Abbreviation: ITT = intent-to-treat.

Note: Only the subset of subjects who were selected to undergo gynecological exams prior to and following tampon use completed the packaging and labeling interview. The packaging and labeling interview was conducted at the Screening/Baseline Visit (Visit 1). Percentages are n/Number of subjects in the ITT Population who belong to the subset of subjects that were selected to undergo gynecological exams and responded to the respective question \*100.

n is the total number of diary entries for each section of the table. N is the number of subjects within each article and within absorbency arm. Reference Listing: 16.2.6.3





# Table 14.2.3 (cont'd.) Summary of Packaging and Labeling Interview Responses ITT Population Gynecological Exam Subset

| Variable | Overa <b>ll</b> |
|---|---|
| Category | (N=XX) |
| Able to correctly identify tampon absorbencies provided in the multipack box | XX |
| Yes | XX (XX,X%) |
| No | XX (XX.X%) |
| Able to correctly identify a regular absorbency wrapped tampon | XX |
| Yes | XX (XX,X%) |
| No | XX (XX.X%) |
| Able to correctly identify a super absorbency wrapped tampon | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Able to correctly identify a super plus absorbency wrapped tampon | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Able to correctly identify the instructions for use from the product insert | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |
| Able to correctly identify the Toxic Shock Syndrome warning from the product insert | XX |
| Yes | XX (XX.X%) |
| No | XX (XX.X%) |

Abbreviation: ITT = intent-to-treat.

Note: Only the subset of subjects who were selected to undergo gynecological exams prior to and following tampon use completed the packaging and labeling interview. The packaging and labeling interview was conducted at the Screening/Baseline Visit (Visit 1). Percentages are n/Number of subjects in the ITT Population who belong to the subset of subjects that were selected to undergo gynecological exams and responded to the given question\*100.

Reference Listing: 16.2.6.3





Table 14.3.1.1
Overall Summary of Adverse Events
Safety Population

Absorbency Arm: Regular

| _ | Before Any Test Article Use | During and Fo <b>ll</b> owing Test<br>Tampon Use | During and Following Reference<br>Tampon Use |
|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 AE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 AE by Severity [1] | | | |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 AE by Relationship [2] | | | |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unlikely | XX (XX,X%) | XX (XX.X%) | XX (XX,X%) |
| Possible | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Probable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Definite | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 AE by Frequency [3] | | | |
| Single | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Intermittent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Continuous | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Subjects with at least 1 SAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; SAE = serious adverse event.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency group\*100. AEs that began prior to insertion of any test article are summarized under Before Any Test Article Use. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use, and AEs that began on or after the date of insertion of first reference tampon are summarized under During and Following Reference Tampon Use. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first reference tampon and prior to date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use. N is the number of subjects within each period and within absorbency arm.

- [1] Subjects are counted only once at the worst severity. If a severity designation is missing, it will be considered as Severe.
- [2] Subjects are counted only once at the strongest possible relationship. If a relationship designation is missing, it will be considered as Definite.
- [3] Subjects are counted only once at the highest possible frequency. If a frequency designation is missing, it will be considered as Continuous. Reference Listing: 16.2.7.1

Programming Note: Repeat for Absorbency Arm: Super.





### Table 14.3.1.2 Adverse Events by System Organ Class and Preferred Term Safety Population

Absorbency Arm: Regular

| Before Any Test Article Use (N=XX) | During and Following Test<br>Tampon Use<br>(N=XX) | During and Following Reference<br>Tampon Use<br>(N=XX) |
|---|---|---|
| XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XX (XX,X%) | XX (XX,X%) | XX (XX,X%) |
| | XX (XX,X%) | XX (XX.X%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XX (XX.X%) | XX (XX.X%) | XX (XX,X%) |
| XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| _ | XX (XX,X%) | Before Any Test Article Use (N=XX) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency group\*100. AEs were coded using MedDRA version 25.1. AEs that began prior to insertion of any test article are summarized under Before Any Test Article Use. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are summarized under During and Following Test Tampon Use, and AEs that began on or after the date of insertion of first reference tampon are summarized under During and Following Reference Tampon Use. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first reference tampon and prior to date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. N is the number of subjects within each article and within absorbency arm.

Reference Listing: 16.2.7.1

Programming Note: Repeat for Absorbency Arm: Super.





Table 14.3.1.3

Adverse Events by System Organ Class, Preferred Term, and Maximum Severity
Safety Population

| System Organ Class | | During and Following Test | During and Following Reference |
|---|---|---|---|
| Preferred Term | Before Any Test Article Use | Tampon Use | Tampon Use |
| Severity | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 AE | XX (XX.X%) | XX (XX.X%) | XX (XX,X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency group\*100. AEs were coded using MedDRA version 25.1. AEs that began prior to insertion of any test article are summarized under Refore Any Test Article Use. For subjects randomized to use the test tampon first. AEs that began on or after the date of

insertion of any test article are summarized under Before Any Test Article Use. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are summarized under During and Following Test Tampon Use, and AEs that began on or after the date of insertion of first reference tampon are summarized under During and Following Reference Tampon Use. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use. Subjects are counted once for each SOC and once for each PT. The severity shown is the greatest severity reported for a particular subject (Severe > Moderate > Mild). AEs with a missing severity were counted as Severe. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. N is the number of subjects within each article and within absorbency arm.

Reference Listing: 16.2.7.1

Programming Note: Repeat for Absorbency Arm: Super.





Table 14.3.1.4

Adverse Events by System Organ Class, Preferred Term, and Maximum Relationship to Study Product Safety Population

| System Organ Class | | During and Following Test | During and Following Reference |
|---|---|---|---|
| Preferred Term | Before Any Test Article Use | Tampon Use | Tampon Use |
| Relationship | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 AE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unlikely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Possible | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| Probable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Definite | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Unlikely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Possible | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Probable | XX (XX.X%) | XX (XX,X%) | XX (XX.X%) |
| Definite | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | | | |
| Not Related | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| Unlikely | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Possible | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Probable | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Definite | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency group\*100. AEs were coded using MedDRA version 25.1. AEs that began prior to insertion of any test article are summarized under Before Any Test Article Use. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are summarized under During and Following Test Tampon Use, and AEs that began on or after the date of insertion of first reference tampon are summarized under During and Following Reference Tampon Use. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use. Subjects are counted once for each SOC and once for each PT. The relationship shown is the greatest relationship reported for a particular subject (Definite > Probable > Possible > Unlikely > Not Related). AEs with a missing relationship were counted as Definite. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by

PT. N is the number of subjects within each article and within absorbency arm. Reference Listing: 16.2.7.1

Programming Note: Repeat for Absorbency Arm: Super.





Table 14.3.1.5

Adverse Events by System Organ Class, Preferred Term, and Maximum Frequency Safety Population

| System Organ Class | | During and Following Test | During and Following Reference |
|---|---|---|---|
| Preferred Term | Before Any Test Article Use | Tampon Use | Tampon Use |
| Frequency | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 AE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Single | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Intermittent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Continuous | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Single | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Intermittent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Continuous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Sing <b>l</b> e | XX (XX,X%) | XX (XX.X%) | XX (XX.X%) |
| Intermittent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Continuous | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Single Single | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Intermittent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Continuous | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities; PT = preferred term; SOC = system organ class.

Note: Percentages are n/Number of subjects in the Safety Population within absorbency group\*100. AEs were coded using MedDRA version 25.1. AEs that began prior to insertion of any test article are summarized under Before Any Test Article Use. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are summarized under During and Following Reference Tampon Use. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first reference tampon and prior to date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Reference Tampon Use, and AEs that began on or after the date of insertion of first test tampon are summarized under During and Following Test Tampon Use. Subjects are counted once for each SOC and once for each PT. The frequency shown is the greatest frequency reported for a particular subject (Continuous > Intermittent > Single). AEs with a missing frequency were counted as Continuous. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. N is the number of subjects within each article and within absorbency arm.

Reference Listing: 16.2.7.1

Programming Note: Repeat for Absorbency Arm: Super.





## Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term Safety Population

Same as shell 14.3.1.2; Programming Note: Replace "Subjects with at least 1 AE" with "Subjects with at least 1 Serious AE".





#### Table 14.3.3.1 Listing of Serious Adverse Events Safety Population

Absorbency Arm: Regular

| Subject<br>ID<br>XXXXXX | Study Period [1] During and Following Test | System Organ Class/ Preferred Term/ Verbatim Term XXXXXXXXXXXX XXXXXXXXXXXX XXXXXXXX | Start Date (Study<br>Day)/ End Date<br>(Study Day)<br>DDMMMYYYY<br>(XX)/<br>DDMMMYYYY<br>(XX) | Severity/ Relationship/ Frequency XXXXXXXX/ XXXXXXXXXXXXXXX | Serious?/<br>Criteria Met<br>Yes/<br>XXXXXXXX | Concomitant<br>medication(s)<br>given? [2]<br>XXX | Outcome/Study<br>Product Action<br>Taken<br>XXXXXXX/<br>XXXXX | Study Product<br>Interruption<br>Start Date<br>(Study Day) /<br>End Date<br>(Study Day)<br>DDMMMYYYY<br>(XX)/<br>DMMMYYYY<br>(XX) | Caused<br>Discontinuation<br>from Study?<br>XX |
|---|---|---|---|---|---|---|---|---|---|
| | Tampon Use During and Following Reference Tampon Use | XXXXXXXXXX<br>XXXXXXXXXXX/<br>XXXXXXXXXX | DDMMMYYYY<br>(XX)/<br>Ongoing | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes/<br>XXXXXXXX | xxx | XXXXXX/<br>XXXXX | (**) | xx |
| | Before Any<br>Test Article<br>Use | XXXXXXXXXX<br>XXXXXXXXXXX/<br>XXXXXXXXXX | DDMMMYYYY (-<br>XX)/<br>DDMMMYYYY<br>(XX) | XXXXXXX/<br>XXXXXXXXXX<br>XXXXXXXXXX | Yes/<br>XXXXXXX | xxx | XXXXXX/<br>XXXXX | | XX |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon). AEs were coded using MedDRA version 25.1. [1] AEs that began prior to insertion of any test article are listed as the Before Any Test Article Use period. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are listed under the During and Following Test Tampon Use period, and AEs that began on or after the date of insertion of first reference tampon are listed under the During and Following Reference Tampon Use period. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first reference tampon and prior to date of insertion of first test tampon are listed under the During and Following Reference Tampon Use period, and AEs that began on or after the date of insertion of first test tampon are listed under the During and Following Test Tampon Use period.

[2] If a concomitant medication was given due to the AE, this will be identified in the prior and concomitant medications listing.

Programming Note: Concatenate all serious criteria marked as Yes with a semicolon. Concatenate all actions taken marked as Yes with a semicolon. If Action Taken, Other is Yes, then concatenate 'Other:' with the text provided in If Other, specify. If no text is provided in If Other, specify, then list 'Other: Not specified'. If no events meet the criteria for display, present "No events are reported." All system organ class and preferred term text should be in proper case. Continue for Absorbency Arm: Super.





# Table 14.3.6.1.1 Gynecological Examination – Visual Assessment Details Safety Population Gynecological Exam Subset

| isit | | |
|-------------------------|-------------|------------------|
| Area Examined | | |
| Assessment | Test Tampon | Reference Tampon |
| Category | (N=XX) | (N=XX) |
| re-Use Visit | | |
| Perineum | | |
| Any Lesions | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Not Done | XX (XX.X%) | XX (XX.X%) |
| Type A Lesions [1] | XX (XX.X%) | XX (XX.X%) |
| Erythema | XX (XX.X%) | XX (XX.X%) |
| Edema | XX (XX.X%) | XX (XX.X%) |
| Coverage of Lesions [2] | | |
| 50% or less | XX (XX,X%) | XX (XX.X%) |
| Greater than 50% | XX (XX.X%) | XX (XX.X%) |
| Type B Lesions [1] | XX (XX.X%) | XX (XX.X%) |
| Petechia | XX (XX.X%) | XX (XX.X%) |
| Ecchymoses | XX (XX.X%) | XX (XX.X%) |
| Coverage of Lesions [2] | , | , |
| 50% or less | XX (XX.X%) | XX (XX.X%) |
| Greater than 50% | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety Population who belong to the subset of subjects that were selected to undergo gynecological exams within tampon type\*100. For the gynecological exam subset, exams were conducted at pre- and post-use visits for each tampon type. Subjects used each tampon type (reference or test) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle. Not Done means that gynecological exam was not done. Subjects XXX,XXX have any lesions found.

- [1] Subjects are counted only once for each type of lesion.
- [2] Subjects are counted only once for the highest coverage lesion recorded for each lesion type.
- n is the number of subjects within each category. N is the number of subjects within each article and within absorbency arm. Reference Listing: 16.2.9.1.1

ū

Programming Note: There will be a pre-use visit and a post-use visit for each tampon type for each subject. Repeat for Absorbency Arm: Super.





# Table 14.3.6.1.1 (cont'd.) Gynecological Examination – Visual Assessment Details Safety Population Gynecological Exam Subset

| Absorbency Arm: Regular | | |
|------------------------------------|-------------|------------------|
| Visit | | |
| Area Examined | | |
| Assessment | Test Tampon | Reference Tampon |
| Category | (N=XX) | (N=XX) |
| Pre-Use Visit | | |
| Perineum (cont'd.) | | |
| Type C Lesions [1] | XX (XX.X%) | XX (XX.X%) |
| Epithelium: Disrupted, superficial | XX (XX.X%) | XX (XX.X%) |
| Epithelium: Disrupted, deep | XX (XX.X%) | XX (XX.X%) |
| Blood vessel: Intact | XX (XX.X%) | XX (XX.X%) |
| Blood vessel: Disrupted | XX (XX.X%) | XX (XX,X%) |
| Peeling | XX (XX.X%) | XX (XX.X%) |
| Abrasion | XX (XX.X%) | XX (XX,X%) |
| Ulceration | XX (XX.X%) | XX (XX.X%) |
| Laceration | XX (XX.X%) | XX (XX.X%) |
| Coverage of Lesions [2] | , | , , |
| 50% or less | XX (XX.X%) | XX (XX.X%) |
| Greater than 50% | XX (XX.X%) | xx (xx.x%) |
| Type D Lesions [1] | XX (XX.X%) | XX (XX.X%) |
| Coverage of Lesions [2] | , | , |
| 50% or less | XX (XX.X%) | XX (XX.X%) |
| Greater than 50% | XX (XX.X%) | XX (XX.X%) |

Repeat for the following areas examined: Vulva, Urethra, Vagina, Cervix; Repeat for the following visit: Post-Use Visit

Note: Percentages are n/Number of subjects in the Safety Population who belong to the subset of subjects that were selected to undergo gynecological exams within tampon type\*100. For the gynecological exam subset, exams were conducted at pre- and post-use visits for each tampon type. Subjects used each tampon type (reference or test) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle.

Programming Note: There will be a pre-use visit and a post-use visit for each tampon type for each subject. Repeat for Absorbency Arm: Super.

<sup>[1]</sup> Subjects are counted only once for each type of lesion.

<sup>[2]</sup> Subjects are counted only once for the highest coverage lesion recorded for each lesion type.

Reference Listing: 16.2.9.1.1





# Table 14.3.6.1.2 Gynecological Examination – Additional Findings Safety Population Gynecological Exam Subset

| /isit<br>Area Examined | Test Tampon | Reference Tampon |
|------------------------------|-------------|------------------|
| Statistic or Category | (N=XX) | (N=XX) |
| Pre-Use Visit | | |
| Vaginal Discharge – Quantity | | |
| Scant | XX (XX.X%) | XX (XX,X%) |
| Small Amount | XX (XX.X%) | XX (XX.X%) |
| Moderate Amount | XX (XX.X%) | XX (XX.X%) |
| Profuse | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |
| Vaginal Discharge – Odor | | |
| Malodorous | XX (XX.X%) | XX (XX.X%) |
| Non-Malodorous | XX (XX.X%) | XX (XX,X%) |
| Missing | XX (XX.X%) | XX (XX X%) |
| Vaginal Discharge – Color | | |
| Clear | XX (XX.X%) | XX (XX.X%) |
| White | XX (XX.X%) | XX (XX.X%) |
| Yellow | XX (XX.X%) | XX (XX.X%) |
| Green | XX (XX.X%) | XX (XX.X%) |
| Red (Bloody) | XX (XX.X%) | XX (XX.X%) |
| Gray | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety Population who belong to the subset of subjects that were selected to undergo gynecological exams within tampon type\*100. For the gynecological exam subset, exams were conducted at pre- and post-use visits for each tampon type. Subjects used each tampon type (reference or test) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle. n is the number of subjects within each category. N is the number of subjects within each article and within absorbency arm.

Subjects XXX,XXX had any abnormal gynecological findings. Subjects XXX,XXX reported any clinically significant gynecological exam result.

Reference Listing: 16.2.9.1.2

Programming Note: There will be a pre-use visit and a post-use visit for each tampon type for each subject. Repeat for Absorbency Arm: Super.





| /isit | T4 T | Defense Tenne |
|---------------------------------|--------------|------------------|
| Area Examined | Test Tampon | Reference Tampon |
| Statistic or Category | (N=XX) | (N=XX) |
| Pre-Use Visit | | |
| Vaginal Discharge – Consistency | | |
| Thin | XX (XX.X%) | XX (XX.X%) |
| Thick | XX (XX.X%) | XX (XX.X%) |
| Variable | XX (XX.X%) | XX (XX.X%) |
| Cottage Cheese Like | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |
| Vaginal pH | | |
| n | XX | XX |
| Mean (SD) | XX,X (XX,XX) | XX.X (XX.XX) |
| Median | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX |
| Suspected Infection | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety Population who belong to the subset of subjects that were selected to undergo gynecological exam within tampon type\*100. For the gynecological exam subset, exams were conducted at pre- and post-use visits for each tampon type. Subjects used each tampon type (reference or test) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle.

Reference Listing: 16.2.9.1.2

Programming Note: There will be a pre-use visit and a post-use visit for each tampon type for each subject. Repeat for Absorbency Arm: Super.





## Table 14.3.6.1.2 (cont'd.) Gynecological Examination – Additional Findings Safety Population Gynecological Exam Subset

| Area Examined | Test Tampon | Reference Tampon |
|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) |
| Pre-Use Visit | | |
| Other Abnormal Findings | | |
| Yes | XX (XX,X%) | XX (XX,X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |
| Gynecological Exam Result Clinically Significant | | |
| Yes | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) |

Note: Percentages are n/Number of subjects in the Safety Population who belong to the subset of subjects that were selected to undergo gynecological exam within tampon type\*100. For the gynecological exam subset, exams were conducted at pre- and post-use visits for each tampon type. Subjects used each tampon type (reference or test) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle.

Reference Listing: 16.2.9.1.2

Programming Note: There will be a pre-use visit and a post-use visit for each tampon type for each subject. Repeat for Absorbency Arm: Super.





### 14.3. Planned Listing Shells

See Figure 3 below.





### **Figure 3: Planned Listing Shells**

Listing 16.2.1.1 Subject Disposition All Subjects

| Arm: XXX | | | | |
|---|---|---|---|---|
| Subject Status | Date of Completion /<br>Discontinuation<br>(Study Day) | Reason for Discontinuation | If Death, Date of Death<br>(Study Day)/<br>Cause of Death | If Lost to Follow-Up,<br>Date of Last Contact (Study Day)/<br>Comment |
| xxxxxxxxxx | DDMMMYYYY (XX) | | | |
| xxxxxxxxxx | DDMMMYYYY (XX) | XXXXXXXXX | | |
| xxxxxx | DDMMMYYYY (XX) | xxxxxxxx | DDMMMYYYY (XX)/<br>XXXXXXXXXX | |
| xxxxxx | DDMMMYYYY (XX) | xxxxxxxx | | DDMMMYYYY (XX)/<br>XXXXXXXXXX |
| | Subject Status XXXXXXXXXX XXXXXXXXXX XXXXXXXXX | Date of Completion / Discontinuation (Study Day) XXXXXXXXXXXX DDMMMYYYY (XX) XXXXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) | Date of Completion / Discontinuation (Study Day) Reason for Discontinuation XXXXXXXXXXX DDMMMYYYY (XX) XXXXXXXXXXX DDMMMYYYY (XX) XXXXXXXXXX XXXXXXXX DDMMMYYYY (XX) XXXXXXXXX | Date of Completion / Discontinuation (Study Day) Subject Status DDMMMYYYY (XX) XXXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) XXXXXXXXX DDMMMYYYY (XX) XXXXXXXXXX DDMMMYYYY (XX) |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

**Programming Note:** If reason for discontinuation is present, concatenate reason for discontinuation with specify text, e.g., "Adverse Event: XXXXX". If a secondary cause of death is listed, concatenate to the primary cause of death with a semicolon. Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





#### Listing 16.2.2.1 Inclusion and Exclusion Criteria All Subjects

| Absorbency A | Arm: XXX | | |
|---|---|---|---|
| Subject ID | Date Screened | Met All Eligibility Criteria? | Criteria Not Met/Reason Not Met |
| xxxxx | DDMMMYYYY | Yes | |
| XXXXX | DDMMMYYYY | Yes | |
| xxxxx | DDMMMYYYY | No | Inclusion #1/XXXXXXXXXXXXXXX; Exclusion #9/XXXXXXXXXXXXX |
| xxxxx | DDMMMYYYY | Yes | |

Programming Note: If there is no "Reason Not Met" included for the corresponding criteria not met, then concatenate the criteria not met with "Reason not given", e.g., "Inclusion #1/Reason not given". If there are multiple criteria met, please list each criteria/reason not met concatenated with a ";". Repeat for Absorbency Arm: Regular and Absorbency Arm: Super. Display screen failures at the end of the listing. For screen failures, the top row will read "Absorbency Arm: Not Assigned (Screen Failures)".





### Listing 16.2.2.2 Protocol Deviations All Subjects

| Absorbency A | Arm: XXX | | | | | |
|---|---|---|---|---|---|---|
| Subject ID | Any Major<br>Protocol<br>Deviations? | Deviation<br>Occurred During a<br>Time Frame? | Deviation Start Date (Study Day)/<br>Deviation End Date (Study Day) | First Visit Impacted/<br>Last Visit Impacted | Protocol Deviation Category | Description |
| xxxxx | No | | | | | |
| xxxxx | Yes | Yes | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXXXXXX/<br>XXXXXXX | xxxxxxxxx | |
| | | No | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXXXXXX/<br>XXXXXXX | xxxxxxxxx | |
| XXXXX | Yes | Yes | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXXXXXX/<br>XXXXXXX | xxxxxxxxx | |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

Programming Note: If "Deviation Occurred During a Time Frame?" is "No" then repeat Deviation Start Date (Study) for Deviation End Date (Study Day) and repeat First Visit Impacted for Last Visit Impacted. If there is text for "Additional Description" (Other than "NA", "N/A" and similar)", then concatenate that text with the text for "Description", e.g., "DESCRIPTION TEXT XXX. ADDITIONAL TEXT." Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





## Listing 16.2.2.3 Reason for Screen Failures Screen Failures

| Subject ID | Failed Date | Met All Eligibility Criteria? | Criteria Not Met/Reason Not Met |
|---|---|---|---|
| XXXXX | DDMMMYYYY | No | Inclusion #4/XXXXXXXXXXXXXXX;<br>Exclusion #2/XXXXXXXXXXXXX |
| XXXXX | DDMMMYYYY | No | Inclusion #1/XXXXXXXXXXXXXXXX;<br>Exclusion #9/XXXXXXXXXXXXX |
| XXXXX | DDMMMYYYY | No | Inclusion #8/XXXXXXXXXXXXXXX; Exclusion #5/XXXXXXXXXXXXX |
| XXXXX | DDMMMYYYY | No | Inclusion #6/XXXXXXXXXXXXXXX;<br>Exclusion #12/XXXXXXXXXXXXX |

Programming Note: If there is no "Reason Not Met" included for the corresponding criteria not met, then concatenate the criteria not met with "Reason not given", e.g., "Inclusion #1/Reason not given". If there are multiple criteria met, please list each criteria/reason not met concatenated with a ";".





#### Listing 16.2.3.1 Analysis Populations All Subjects

Absorbency Arm: XXX

| | | Randomization | ation Analysis Populations | | _ | | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Date | Number | Tampon Used<br>First | Part of<br>Subset? [1] | ITT [2] | Safety [3] | MITT [4] | Primary Reason(s) for Exclusion |
| xxxxxx | DDMMMYYYY | XXXX | xxxxxxx | xxxxxxx | Yes | No | No | Safety: Subject did not insert any tampons. |
| XXXXXX | DDMMMYYYY | XXXX | XXXXX | XXXXX | Yes | Yes | Yes | |
| XXXXXX | DDMMMYYYY | XXXX | xxxxxxx | XXXXXXX | Yes | Yes | No | MITT: Subject did not return any tampons that could be assessed for elongation. |
| xxxxx | DDMMMYYYY | xxxx | XXXXX | XXXXXXX | No | No | No | ITT: Subject was not randomized. |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon; CS = super absorbency reference tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tam ITT = intent-to-treat; MITT = modified intent-to-treat.

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.

<sup>[1]</sup> A subset of subjects were selected to undergo gynecological exams prior to and following tampon use. In addition, this subset of subjects completed the packaging and labeling interview at the Screening/Baseline Visit (Visit 1).

<sup>[2]</sup> The ITT Population includes all subjects randomized into the study.

<sup>[3]</sup> The Safety Population includes all ITT subjects who insert at least 1 tampon.

<sup>[4]</sup> The MITT Population includes all subjects in the Safety population who have no major protocol deviations and return at least 1 tampon that can be assessed for elongation.





#### Listing 16.2.4.1 Subject Consent and Demographics All Subjects

| Absorbency | Arm: XXX Date Informed | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject ID | Consent Version | Protocol Version | Date of Birth | Age<br>(years) | Sex | Ethnicity | Race |
| xxxxxx | DDMMMYYYY/<br>XXXXXXXXXXX | xxxxxxxx | DDMMMYYYY | XX | Female | xxxxxx | xxxxxx |
| xxxxxx | DDMMMYYYY/<br>XXXXXXXXXXX | xxxxxxxx | DDMMMYYYY | XX | Female | xxxxxx | XXXXXX |
| xxxxxx | DDMMMYYYY/<br>XXXXXXXXXXX | xxxxxxxx | DDMMMYYYY | XX | Unknown | xxxxxx | xxxxx |
| xxxxxx | DDMMMYYYY/<br>XXXXXXXXXXX | xxxxxxxx | DDMMMYYYY | XX | Female | xxxxxx | xxxxxx |
| xxxxxx | DDMMMYYYY/<br>XXXXXXXXXXX | xxxxxxxx | DDMMMYYYY | XX | Undifferentiated | XXXXXX | XXXXXX |

Programming Note: If multiple races are selected, then concatenate all selected races using a semicolon. Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





Listing 16.2.4.2 Medical History All Subjects

Absorbency Arm: XXX

| Subject ID | Any Medical<br>History<br>Reported? | Date Medical<br>History Collected<br>(Study Day) | Category/<br>Verbatim Term | Start Date (Study Day)/<br>End Date (Study Day) | Medical History<br>Disease/Condition<br>Under Control? |
|---|---|---|---|---|---|
| xxxxxx | Yes | DDMMMYYYY<br>(XX) | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | Yes |
| | | | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXXX | -MMMYYYY /<br>Ongoing | No |
| xxxxxx | Yes | DDMMMYYYY<br>(XX) | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | Yes |
| | | | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | -MMMYYYY /<br>Ongoing | Yes |

Abbreviation: MedDRA = Medical Dictionary for Regulatory Activities.

Note: At the Screening/Baseline Visit (Visit 1), subjects were asked to report any previously ongoing or current medical conditions or procedures that had occurred within 3 months prior to study entry. Medical history was coded using MedDRA version 25.1. Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

Programming Note: If medical history is ongoing, denote with "Ongoing" rather than the end date. Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





### Listing 16.2.4.3 Tampon Use Questionnaire All Subjects

Absorbency Arm: XXX

| Subject ID | Study Visit | Date Completed<br>(Study Day) | Assessment | Result |
|---|---|---|---|---|
| XXXXX | xxxxxxx | DDMMMYYYY (XX) | How many total tampons do you typically use during your period? | xxx |
| | | | What tampon absorbency do you use most often? | XXX |
| | | | Are you willing to use only regular absorbency tampons during your participation in the study, if needed and if you qualify? | XXX |
| | | | Are you willing to use only super absorbency tampons during your participation in the study, if needed and if you qualify? | XXX |
| XXXXX | xxxxxxx | DDMMMYYYY (XX) | How many total tampons do you typically use during your period? | XXX |
| | | ` ' | What tampon absorbency do you use most often? | XXX |
| | | | Are you willing to use only regular absorbency tampons during your participation in the study, if needed and if you qualify? | XXX |
| | | | Are you willing to use only super absorbency tampons during your participation in the study, if needed and if you qualify? | XXX |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

**Programming Note:** If the response for "What tampon absorbency do you use the most?" is "I use approximately equal numbers of 2 or more absorbency tampons" then please concatenate the result with the tampons selected, e.g., "I use approximately equal numbers of 2 or more absorbency tampons: Light; Regular". Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





### Listing 16.2.5.1 Test Article and Diary Dispensation and Diary Training All Subjects

Absorbency Arm: XXX

| Subject ID | Study Visit | Test Article and<br>Diary Dispensation<br>Completed? | Diary Training Performed?/<br>Reason Not Performed | Diary<br>Number | Lot Number of<br>Tampons<br>Dispensed | Tampon Code<br>Dispensed | Dispensation Date<br>(Study Day) |
|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXXXX | Yes | Yes | XX | xx | XX | DDMMMYYYY (XX) |
| | xxxxxxxx | Yes | No/<br>XXXXXXXXXXXXXX | XX | XX | XX | DDMMMYYYY (XX) |
| XXXXX | XXXXXXXX | Yes | Yes | XX | XX | XX | DDMMMYYYY (XX) |
| | xxxxxxxx | No | No/<br>XXXXXXXXXXXXXXXX | XX | XX | XX | DDMMMYYYY (XX) |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon,

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





Listing 16.2.5.2 Diary Review Safety Population

Absorbency Arm: XXX

| Subject ID | Study Visit | Date Returned<br>(Study Day) | Diary<br>Number | Tampon<br>Code | Diary Entry for Each<br>Tampon Used? | Are A <b>ll</b> Diary Entries Accurate and Complete? | Were All Discrepancies Addressed and Corrected with Subject? |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxx | DDMMMYYYY (XX) | 1 | xx | Yes | Yes | |
| | xxxxxxxx | DDMMMYYYY (XX) | 2 | xx | No | No | No; XXXXXXXXXXXXXXX |
| XXXXX | xxxxxxxx | DDMMMYYYY (XX) | 1 | XX | Yes | No | Yes |
| | xxxxxxxx | DDMMMYYYY (XX) | 2 | XX | Yes | Yes | |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).





### Listing 16.2.6.1 Tampon Integrity Assessment Safety Population

Absorbency Arm: XXX

| Subject ID | Study Visit | Assessment<br>Performed?/<br>Reason Not<br>Performed | Assessment<br>Date (Study<br>Day) | Number of<br>Used<br>Tampons<br>Returned | Number of<br>Unused<br>Tampons<br>Returned | Menstrual<br>Cycle | Tampon<br>Code<br>Returned | Tampon<br>Number | Length of<br>Elongation<br>(mm) | Elongated [1]? | Picture<br>Taken of<br>Tampon? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | No/<br>XXXXXXXXXXX | | | | | | | | | |
| XXXXXX | xxxxxx | Yes | DDMMMYYYY<br>(XX) | XX | XX | XX | XX | XX | XX | No | Yes |
| | | | | | | XX | XX | XX | XX | No | Yes |
| | | | | | | XX | XX | XX | XX | Yes | Yes |
| | | | | | | XX | XX | XX | XX | XX | No |
| | | | | | | XX | XX | XX | XX | XX | XX |
| | | | | | | XX | XX | XX | XX | XX | XX |
| | | | | | | XX | XX | XX | XX | XX | XX |
| | | | | | | XX | XX | XX | XX | XX | XX |
| | xxxxx | Yes | DDMMMYYYY<br>(XX) | xx | xx | XX | XX | XX | xx | XX | XX |
| | | | (, , , | | | XX | XX | XX | XX | XX | XX |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon. Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

[1] Any used tampon with a measurement of elongation >10 mm was considered elongated.

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





### Listing 16.2.6.2.1 Individual Tampon Entry Diary Responses Safety Population

Absorbency Arm: XXX

| Subject | | Diary | Tampon | Entry | Date/Time (Study Day) | Date/Time (Study Day) | Able to<br>Remove | White Area<br>Remaining on | Flow When<br>Using | |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Study Visit | Number | Code | Number | Tampon Inserted | Tampon Removed | Tampon? | Tampon? | Tampon? | Comments |
| xxxxx | xxxxxx | 1 | XX | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | xx | xxxxxx | xxxx | |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | XXXXXX |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | XXXXXX |
| | xxxxxx | 2 | XX | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | xxxxxx | xxxx | |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | XXXXXX |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | |
| xxxxx | xxxxxx | 1 | XX | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | xxxxx | xxxx | |
| | | | | XX | DDMMMYYYY/HH:MM<br>(XX) | DDMMMYYYY/HH:MM<br>(XX) | XX | XXXXXX | XXXX | XXXXXX |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon. Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

**Programming Note:** Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





### Listing 16.2.6.2.2 Diary Responses Following Last Tampon Use Safety Population

Absorbency Arm: XXX

| Subject<br>ID | Study Visit | Diary<br>Number | Tampon<br>Code | Assessment | Response |
|---|---|---|---|---|---|
| xxxxx | XXXXXXX | 1 | XX | Were you able to open the box to retrieve the wrapped tampons? Were you able to open each tampon wrapper? Were each of the tampons clean prior to using them? Were you able to insert each tampon using the applicator? | Yes<br>Yes<br>Yes<br>Yes |
| | xxxxxx | 2 | XX | Were you able to open the box to retrieve the wrapped tampons? Were you able to open each tampon wrapper? Were each of the tampons clean prior to using them? Were you able to insert each tampon using the applicator? | Yes<br>No; XXXXXXXXXX<br>Yes<br>No |
| xxxxx | XXXXXXX | 1 | XX | Were you able to open the box to retrieve the wrapped tampons? Were you able to open each tampon wrapper? Were each of the tampons clean prior to using them? Were you able to insert each tampon using the applicator? | Yes<br>Yes<br>Yes<br>Yes |
| | xxxxxx | | | | |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon.

Programming Note: If the response for any of the assessments "Were you able to open the box to retrieve the wrapped tampons?", "Were you able to open each tampon wrapper?", or "Were each of the tampons clean prior to using them?" is "No" then concatenate the text from the corresponding "If no, please explain in detail", e.g., "No; XXXXXXXXXX". If the response for the assessment "Were you able to insert each tampon using the applicator?" is "No", then keep it as 'No' without the details.

Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.





### Listing 16.2.6.2.3 Reason for Not Inserting the Tampon Using the Applicator Safety Population

Absorbency Arm: XXX

| Subject<br>ID | Study<br>Visit | Diary<br>Number | Tampon<br>Code | Reason | Explain in Detail, Why You Were Not Able to Insert Each<br>Tampon Using the Applicator | Comments |
|---|---|---|---|---|---|---|
| xxxxx | xxxxxx | 1 | XX | XXXX; XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxx |
| | xxxxxx | 2 | XX | XXXX; XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXX |
| XXXXX | xxxxxx | 1 | XX | XXXX; XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXX |
| | xxxxxx | | | | | |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon.

**Programming Note:** Repeat for Absorbency Arm: Regular and Absorbency Arm: Super. In case of several reasons, please concatenate them by ";".





### Listing 16.2.6.3 Packaging and Labeling Interview Gynecological Exam Subset

| Absorbency | Arm: XXX | Assessment Performed?/ | Assessment Date | Interviewer | | |
|---|---|---|---|---|---|---|
| Subject ID | Study Visit | Reason Not Done | (Study Day) | Initials | Assessment | Response |
| xxxxx | XXXXXXX | No/XXXXXXX | | | | |
| XXXXX | xxxxxx | Yes | DDMMMYYYY (XX) | xx | What tampon absorbency or absorbencies are provided in this box? / Was subject able to identify the correct information? | XXXX/Yes |
| | | | | | Show me where you found that information / Was subject able to identify the correct information? | NA |
| | | | | | Can you show me the tampon absorbency ranges for the entire line of products on the box? | XX |
| | | | | | Can you show me the Toxic Shock Syndrome warning on the box? | XX |
| | | | | | Can you show me on the bow where the information is that states how long you should use a tampon? | XX |
| | | | | | What tampon absorbency or absorbencies are provided in this box? / Was subject able to identify the correct information? | XXXX/No |
| | | | | | Show me where you found that information / Was subject able to identify the correct information? | XX/Yes |
| | | | | | What tampon absorbency or absorbencies are provided in this box? / Was subject able to identify the correct information? | XXXX/No |
| | | | | | Show me where you found that information / Was subject able to identify the correct information? | XX/Yes |
| | | | | | What tampon absorbency or absorbencies are provided in this box? / Was subject able to identify the correct information? Show me where you found that information / Was subject able to identify the correct information? | XXX/ |
| | | | | | Can you identify a regular absorbency wrapped tampon? | XX |
| | | | | | Can you identify a super absorbency wrapped tampon? | XX |
| | | | | | Can you identify a super plus absorbency wrapped tampon? | XX |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super.

product insert?

Can you show me the instructions for use on the product insert?

Can you show me the Toxic Shock Syndrome warning on the

AD-ST-33.06 Effective date: 12-Nov-2020

XX

XX





Study Product

Listing 16.2.7.1 Adverse Events All Subjects

Absorbency Arm: XXX

| Subject<br>ID<br>XXXXXX | Study Pr<br>Period [1] During and XXX<br>Following XX | stem Organ<br>ss/<br>referred Term/<br>Verbatim Term<br>XXXXXXXXX<br>XXXXXXXXXXXXXXXXXXXXXXXXXX | Start Date (Study<br>Day)/ End Date<br>(Study Day)<br>DDMMMYYYY<br>(XX)/<br>DDMMMYYYY<br>(XX) | Severity/ Relationship/ Frequency XXXXXXX/ XXXXXXXXXXXXXXXXXXXXXXXXXXXX | Serious?/<br>Criteria Met<br>Yes/<br>XXXXXXXX | Concomitant<br>medication(s)<br>given? [2]<br>XXX | Outcome/Study<br>Product Action<br>Taken<br>XXXXXXX/<br>XXXXX | Interruption Start Date (Study Day) / End Date (Study Day) DDMMMYYYY (XX)/ DMMMYYYY (XX) | Caused<br>Discontinuation<br>from Study?<br>XX |
|---|---|---|---|---|---|---|---|---|---|
| | During and XXX | XXXXXXXX<br>XXXXXXXXXX/<br>XXXXXXXXXX | DDMMMYYYY<br>(XX)/<br>Ongoing | XXXXXXX/<br>XXXXXXXXXX<br>XXXXXXXXXX | No | XXX | XXXXXX/<br>XXXXX | | XX |
| <b>XXXXXX</b> | • | XXXXXXXX<br>XXXXXXXXXX<br>XXXXXXXXX | DDMMMYYYY (-<br>XX)/<br>DDMMMYYYY<br>(XX) | XXXXXXX/<br>XXXXXXXXXX<br>XXXXXXXXXX | No | xxx | XXXXXX/<br>XXXXX | | XX |
| | | | DDMMMYYYY | | | | XXXXX | | |

Abbreviations: AE = adverse event; MedDRA = Medical Dictionary for Regulatory Activities.

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon). AEs were coded using MedDRA version 25.1. [1] AEs that began prior to insertion of any test article are listed as the Before Any Test Article Use period. For subjects randomized to use the test tampon first, AEs that began on or after the date of insertion of first test tampon and prior to date of insertion of first reference tampon are listed under the During and Following Test Tampon Use period, and AEs that began on or after the date of insertion of first reference tampon are listed under the During and Following Reference Tampon Use period. For subjects randomized to use the reference tampon first, AEs that began on or after the date of insertion of first reference tampon and prior to date of insertion of first test tampon are listed under the During and Following Reference Tampon Use period, and AEs that began on or after the date of insertion of first test tampon are listed under the During and Following Test Tampon Use period.

[2] If a concomitant medication was given due to the AE, this will be identified in the prior and concomitant medications listing.

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super





### Listing 16.2.9.1.1 Gynecological Examination – Visual Assessment Details Gynecological Exam Subset

Absorbency Arm: XXX

| Subject<br><b>I</b> D | Study Visit | Exam Performed?/<br>Reason Not Performed | Exam Date<br>(Study Day) | Clinically<br>Significant<br>Result? | Area<br>Examined | Lesions?/<br>Type/<br>Coverage (%) | Comment |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxx | Yes | DDMMMYYYY<br>(XX) | No | Perineum | No | |
| | | | , | | Vulva | Yes/<br>Type A; Edema<br>50 or <b>l</b> ess | XXXXXXXX |
| | | | | | Urethra<br>Vagina | No<br>Yes<br>Type C; Disrupted, Deep; Intact;<br>Peeling | |
| | | | | | Cervix | No | |
| | XXXXXXX | No/<br>XXXXXXXXXXXXXXXXXX | | | | | |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon). For the subset of subjects that were selected to undergo gynecological examinations prior to and following tampon use, gynecological exams were conducted at pre-use visits and post-use visits for each test article type. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle.

**Programming Note:** The study visits will include the following: "Pre-test tampon use visit", "Post-test tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit", "Pre-reference tampon use visit", "Pre-reference tampon use visit", "Pre-reference tampon use visit", "Pre-reference tampon use visit", and "Post-reference tampon use visit" and "Post-reference t





Absorbency Arm: XXX

| Subject<br><b>I</b> D | Study Visit | Exam Performed?/<br>Reason Not Performed | Exam Date<br>(Study Day) | Vaginal Discharge Quantity/<br>Odor/<br>Color/<br>Consistency | Vagina <b>l</b><br>pH | Suspected Infection? | Other<br>Abnormal<br>Findings? | Clinically<br>Significant<br>Result? |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxx | Yes | DDMMMYYYY<br>(XX) | XXXXXXXX/<br>XXXXXX/<br>XXXXXXXX/<br>XXXXXXXXXX | xx | No | No | No |
| | XXXXXXX | Yes | DDMMMYYYY<br>(XX) | XXXXXXXX/<br>XXXXXXX/<br>XXXXXXXX/<br>XXXXXXXXXX | XX | Yes | No | Yes |
| | xxxxxxx | No/<br>XXXXXXXXXXXXXXXXXX | | | | | | |
| | xxxxxxx | Yes | DDMMMYYYY<br>(XX) | XXXXXXXX/<br>XXXXXX/<br>XXXXXXXX/<br>XXXXXXXXXX | xx | No | Yes; XXXXXX | No |
| xxxxx | xxxxxxx | No/<br>XXXXXXXXXXXXXXXXXX | | | | | | |

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon). For the subset of subjects that were selected to undergo gynecological examinations prior to and following tampon use, gynecological exams were conducted at pre-use visits and post-use visits for each test article type. Subjects used each test article type (reference or test tampon) over the course of one menstrual cycle. Pre-use visits were conducted within 72 hours prior to expected menstruation and post-use visits were conducted within 72 hours following the last tampon use for that menstrual cycle.

**Programming Note:** The study visits will include the following: "Pre-test tampon use visit", "Post-test tampon use visit", "Pre-reference tam





### Listing 16.2.9.2 Prior and Concomitant Medications All Subjects

| | Any<br>Medications | Prior or | ATC Class (Level 4)/<br>Preferred Term/ | | Start Date (Study Day)/ | | Route/ |
|---|---|---|---|---|---|---|---|
| Subject ID | Reported? | Concomitant [1] | Medication or Therapy | Indication | End Date (Study Day) | Dose (Unit) | Frequency |
| XXXXX | Yes | XXX | XXXXX/<br>XXXXXXXXX/<br>XXXXXXXXXX | XXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX (XXX) | XXXXXXX/<br>XXXXXXX |
| | | XXX; XXX | XXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXX | -MMMYYYY/<br>Ongoing | XXX (XXX) | XXXXXXXX/<br>XXXXXXX |
| | | XXX | XXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX (XXX) | XXXXXXXX/<br>XXXXXXX |

Abbreviations: ATC = Anatomical Therapeutic Chemical Classification System; WHO-DD = World Health Organization Drug Dictionary.

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon). Medications were coded using WHO-DD Enhanced B3 (September 2022).

[1] Prior medications are all medications that were started before the first insertion of the test article. Concomitant medications are all medications that were started after the first insertion of the test article or were continuing after the first insertion of the test article. If a medication starts before the first insertion of the test article and continues after the first insertion of the test article it is considered both prior and concomitant.

Programming Note: If Route, or Frequency is "Other", display "If Other, specify" text only (i.e., do not display "Other: XXXXXX" but just "XXXXXX"). Sort by subject, start date, end date, ATC Level 4 & Preferred Term. Repeat for Absorbency Arm: Regular and Absorbency Arm: Super





### Listing 16.2.9.3 Product Complaints All Subjects

Absorbency Arm: XXX

| Subject ID | Any Product<br>Complaints<br>Reported? [1] | Issue/Problem Date (Study<br>Day) | Product Code | Complaint Description | Device Available to be Examined? |
|---|---|---|---|---|---|
| xxxxx | Yes | DDMMMYYYY (XX)<br>DDMMMYYYY (XX) | XX<br>XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | No<br>Yes |
| xxxxx | No | | | | |
| XXXXXX | Yes | DDMMMYYYY (XX) | XX | xxxxxxxxxxxxx | Yes |

Abbreviations: BR = regular absorbency test tampon; BS = super absorbency test tampon; CR = regular absorbency reference tampon; CS = super absorbency reference tampon.

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

[1] Includes product complaints reported that were not previously captured in the subject diary or as an adverse event.

Programming Note: Repeat for Absorbency Arm: Regular and Absorbency Arm: Super





#### Listing 16.2.10.1 COVID-19 Impact Assessment All Subjects

| Absorbend<br>Subject<br>ID | cy Arm: XXX Subject Affected by COVID- 19? | Visit<br>Impacted | Visit Type<br>Adjustment | Visit Date<br>(Study Day) | Efficacy<br>Assessments<br>Missed? | Safety<br>Assessments<br>Missed? | Early Termination<br>Reason, if attributable<br>to COVID-19 | Comments |
|---|---|---|---|---|---|---|---|---|
| XXXXX | Yes | XXXXX | XXXX | DDMMMYYYY<br>(XX) | xxx | XXX | | XXXXXXX |
| XXXXX | Yes | XXXXX | XXXX; XXXX | DDMMMYYYY<br>(XX) | XX | XXX | XXXXXX | |
| xxxxx | No | | | | | | | |

Abbreviation: COVID-19 = novel coronavirus disease-2019.

Note: Study day is calculated relative to the date of first insertion of study product (either test or reference tampon).

**Programming Note:** If more than once visit type adjustment is selected, then concatenate all selected with a semicolon. If visit type adjustment "Other" is selected, or if "ET reason (if attributable to COVID-19)" is "Other", then display "Other, specify" text only (i.e., do not display "Other: XXXXXXX" but just "XXXXXX"). Repeat for Absorbency Arm: Regular and Absorbency Arm: Super